CLINICAL TRIAL: NCT04719364
Title: A Cross-Sectional Survey of PrEP Awareness, Barriers and Facilitators for PrEP Uptake, and the Impact of Dosing Mechanisms on Willingness to Take PrEP Among MSM Indicated for PrEP Use in Philadelphia
Brief Title: PrEP Awareness, Barriers and Facilitators for PrEP Uptake, and Dosing Mechanisms on Willingness to Take PrEP Among MSM
Acronym: MSM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Drexel University (Other)
Collaborators: Temple University (Other)
Responsible Party: Principal Investigator, Seth Welles, Professor of Epidemiology, Drexel University
Other Study IDs: 480121
Record Dates: First submitted 2020-11-09; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: PrEP; Discrimination, Racial; Stigma, Social
Keywords: PrEP; MSM; Barriers; Facilitators; Discrimination
MeSH Terms: conditions — Racism; Social Stigma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Focus Groups: 10 black, 10 Latinx, and 10 white MSM will be recuited in this focus group 'cohort'
- Quantitative Survey Group: Cross-sectional group of 100 black, 100 Latinx, and 100 white MSM

SUMMARY:
The investigators are conducting a one and one-half year mixed-methods study to evaluate self-reported sexual risk, knowledge and barriers/facilitators of PrEP use, and preferences of oral, injectable, and implantable PrEP treatment modalities-as a function of race and age, and experience with intersectional discrimination. The first qualitative phase of our study would be conducted over the first eight months, followed by a quantitative phase that will collect data via online cross-sectional survey over the remaining ten months.

DETAILED DESCRIPTION:
This mixed-methods project will evaluate PrEP awareness and potential impact of new dosing strategies/modalities on PrEP uptake among men who have sex with men (MSM)-the target group at highest risk for infection and at highest priority for PrEP use based on high risk sexual behaviors (condomless anal intercourse). The proposed project utilizes both qualitative analysis of focus group data from MSM study participants, as well as quantitative analysis of results from a survey informed by results of the qualitative phase of our project. It should be noted that while the investigators will target a racially diverse MSM study population, participation in our study may include MSM who also inject drugs (MSM-PWID) who express interest in study participation.

The investigators propose a one and one-half year mixed-methods study to evaluate self-reported sexual risk, knowledge and barriers/facilitators of PrEP use, and preferences of oral, injectable, and implantable PrEP treatment modalities-as a function of race and age, and experience with intersectional discrimination. The first qualitative phase of our study would be conducted over the first eight months, followed by a quantitative phase that will collect data via online cross-sectional survey over the remaining ten months.

Recruitment for both qualitative and quantitative parts of our project will occur through events sponsored by the Philly Ballroom Community, freeHIVTest.Net, GALAEI and COLOURS (CBOs), and Drexel's HIV Clinical Center, the Partnership Comprehensive Care Practice. For our quantitative survey, the investigators plan to enhance our recruitment using online social media sites that especially target BMSM and HLMSM, and Google Words-the investigators will display links to our study that will enable recruitment.

For qualitative work, the investigators plan to conduct six focus groups of 5 MSM each (total = 30 participants), each restricted by race and age (Black, White, or Hispanic/Latino (either Black or White) and age (18-39 yrs. of age and > 40 yrs. of age). Four to six focus groups are usually recommended to reach saturation. Given probable cultural and age-specific differences of PrEP awareness and knowledge, as well as barriers or facilitators, and preference for specific treatment modalities, the investigators plan to restrict group participation by race and age as outlined above.

Data collected from the 30 focus group participants will be analyzed using standard qualitative analytic approaches (Months 7-8). Drexel University's Dornsife School of Public Health have available a wide range of qualitative data analysis software and strategies for more sophisticated coding, retrieval, and concept development of the information collected in the focus groups. The investigators will utilize standard qualitative techniques, including inductive code identification and development and associated documentation through marginal remarks and memos. Inductive coding ("open coding") involves a data-based approach to the identification of key themes (codes). This approach encourages a conceptualization and organizational framework of the data from a grounded perspective. NVivo, a system for the management, interpretation and analysis of qualitative data, will be used in this process. Results from the qualitative phase of our project will be used to inform/add to the content of our study instrument to collect data during the second, quantitative phase of our project. For the quantitative, cross-sectional survey, the investigators plan to enroll equal numbers of White, Black, and Hispanic/Latino MSM (100 members per racial/ethnic group, for a total of 300 participants).

The study design for this quantitative phase will be cross-sectional, with analysis conducted from a sample of 300 PrEP eligible study participants. The investigators plan to enroll a racially and ethnically diverse study population with 1/3 each White non-Hispanics, Black non-Hispanics, and Hispanic/Latinos. Participants will be recruited in-person at our local CBOs and online. Enrollment and survey conduct will occur at CBO sites and at Drexel's Partnership Comprehensive Care Clinic, as described above. It should be noted that participants in the qualitative phase of our study will be ineligible to participate in the quantitative phase of the study.

Collection of Survey Data. Study participants will use online audio-assisted Red Cap surveys to provide information about demographics, recent sexual risk behaviors, awareness and knowledge concerning PrEP, barriers and facilitators of PrEP use, preference for treatment modalities, and experiences with discrimination. Collection of data will be facilitated by staff at CBO sites, who will log participants onto our study survey data collection site, and who will be available to answer questions/provide clarification as needed. Surveys will be offered in both English and Spanish. The use of audio-assisted self-interviewing is particularly appropriate for collecting data from participants with limited literacy and provides a sense of confidentiality to decrease possibility of prevarication.

Survey Items

Demographics. Survey items will include: Race/ethnicity (White, Black, Hispanic/Latino), age (continuous), education level (less than high school, high school graduate, some college courses or 2 year degree, 4 year college graduate, graduate school courses or degree), employment status, annual income, and self-identified sexual orientation, and perceived need to not disclose/hide one's gay/bi/MSM identity.

Sexual Behaviors. Behavioral data will include 60 day recall of number of men and women with whom participants have had anal or vaginal sex (as appropriate for partners' gender/sex), and for partners with whom participants had anal or vaginal sex: consistency of condom use with partners for whom HIV status was unknown or if partners were HIV-positive; consistency of condom use with partners for whom HIV status known and were HIV-negative; and whether participants have been diagnosed with bacterial STIs within the recall period.

Awareness of PrEP. Survey items concerning awareness of PrEP will be taken from the National HIV Behavioral Risk Surveillance System (NHBS). Survey items will be adapted from national survey questions, and well as questions specific to Philadelphia (see draft study instrument in Appendix). Essentially, participants will be asked whether they have heard of PrEP or Truvada (by name), or if they have heard of medication that would prevent HIV infection if taken daily, or if they have heard of medication (PEP) that is taken after high-risk sexual contact (event-driven regimen). Participants will also be asked if they would reduce use of condoms for anal intercourse and increase the number of sexual partners if they were to take PrEP.

Barriers and Facilitators of PrEP Use. Survey items will be adapted from the NHBS and previously published work by Golub and colleagues (2013) concerning perceived barriers and facilitators of PrEP. Barriers to PrEP use will include: Not being at risk for HIV, not providing full protection from HIV infection, short-term side effects, long-term health effects, stigma/embarrassment around using PrEP, and being too expensive for me/no insurance. Facilitators of PrEP use will include: Being at risk for HIV infection, PrEP will protect from HIV, PrEP will simplify having sex with no need to use condoms, PrEP will simplify having sex with no need to discuss safe sex or HIV status, PrEP is available at no cost to me, I could get ready access to support services (HIV/STI testing and access to sexual health/care monitoring).

Preference for Specific Treatment Modalities. This survey will include items concerning likelihood of using PrEP based on different treatment availability: oral daily dosing, monthly injectable dosing, and yearly implantable dosing of PrEP. A five-point Likert-like scale will be used for each of these, ranging from 'Not at all likely' to 'Fully likely. For those who respond with being 'Somewhat likely' or Fully likely' to used PrEP for each dosing modality, the investigators will ask follow-up questions concerning reasons for higher acceptability including convenience and discretion when non-disclosure of PrEP use is desired.

Experiences with Intersectional Discrimination. The investigators will adapt a newly published, intersectional discrimination scale developed by Scheim and Bauer (2019) that measures experiences with and anticipation of discrimination "because of who patients are", capturing multiple minority identities-including being Black or Hispanic/Latino and being a MSM. In our case, the investigators will use the scale to measure intersectional discrimination in our study population and compare levels (continuous) between specific categories-being BMSM and 18-39 yrs. of age, BMSM > 40 yrs. of age, HLMSM and 18-39 yrs. of age, HLMSM > 40 yrs. of age, WMSM and 18-39 yrs. of age, and WMSM > 40 yrs. of age.

Planned Data Analysis

Descriptive Analysis. Descriptive analysis will be performed using data fields outlined and listed above. For binary or categorical variables, proportion of study participants was given responses will be listed for the entire sample, and proportions will be stratified by race and age as described above. Thus the investigators initially plan to summarize demographics of our sample, including age, race, level of education, whether or not participants are employed, income levels, and self-reported sexual orientation. The investigators will then measure these rates by race and age, comparing differences in proportions across racial/ethnic and age groups by chi-square tests or Fisher's exact tests if data are sparse. For each data field, results will be presented as proportion reporting response options by subgroup, with p-values associated with statistical testing. The convention of p-values < 0.05 as criteria for statistical significance will be utilized for analysis. For variables that are measured continuously, the investigators will use either Student's t-tests (for normally distributed data) or nonparametric methods such as Wilcoxon rank sum tests are not normally distributed data. For each data field median values will be presented along with associated 25%-75% interquartile ranges. Again, p-values will be given for subgroup comparisons.

The investigators plan to test for differences of distributions/levels of sexual behaviors including frequency of condomless anal intercourse, awareness of PrEP, barriers and facilitators of PrEP use, preference for specific PrEP treatment modalities, and experiences with discrimination between subgroups.

Regression Analysis. Subsequently, the investigators will conduct univariate and multivariate regression to identify whether beliefs concerning one's HIV risk, frequencies of sexual behaviors, and level of experience with discrimination (all potential explanatory variables) are associated with awareness PrEP (yes/no), level of knowledge of PrEP effectiveness (high vs. lower), report of specific barriers and facilitators of PrEP use (yes/no), and preference for injectable or implantable PrEP treatment modalities-all dependent or outcome variables.

For each explanatory variable the investigators will estimate outcome variable prevalence ratios using PROC GENMOD (log-linked binomial model) or PROC LOGISTIC (logistic models). The investigators will report unadjusted prevalence ratios with associated 95% confidence intervals and p-values. Ultimately, multiple regression will be used to evaluate estimates of outcome prevalence ratios for explanatory variables, adjusted for confounders that are identified vis-à-vis descriptive analysis and univariate regression. Standard criteria to assess confounding will be used, including a 10% change in the magnitude of association of the independent variables with the various outcome variables.

To identify potential effect modification, stratified analysis (by race/ethnicity, and age) will be conducted, and Wald tests to evaluate homogeneity will be used to test for differences of stratum-specific odds ratios.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifying as gay, bisexual or a man who has sex with men (MSM)
* Being at least 18 years of age; 3) self-reporting as being HIV-negative
* Having had anal intercourse with a man in the past six months
* Not in a monogamous partnership with a recently tested, HIV-negative man AND at least one of the following: Any anal sex without condoms (receptive or insertive) in past 6 months or having been diagnosed with a bacterial STI (syphilis, gonorrhea, or chlamydia) in past 6 months.

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — cis Male
Study Population: The proposed mixed methods study will evaluate PrEP awareness, barriers and facilitators of uptake, and preference for monthly injectable and annual implantable PrEP versus daily oral medication in a diverse racial/ethnic sample of men who have sex with men (MSM). Specifically, we plan to recruit sufficient numbers (n=300 total) of black MSM (n=100) and Hispanic/Latino MSM (n=100), as well as non-Hispanic/Latino White men (n=100) (at least 18 years of age) to enable our team to evaluate disparities concerning PrEP awareness and knowledge, as well as potential preferences for specific treatment modalities.
Sampling Method: Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
condomless anal intercourse | Baseline
  frequency of condomless intercourse with other men
Awareness of PrEP | Baseline
  Survey item adapted from the NHBS-- yes/no
Likelihood of daily PrEP use | Baseline
  5-point Likert scale measuring likelihood of using daily oral PrEP if freely available and covered by insurance
Barriers to PrEP use | Baseline
  6-item checklist of barriers as previously reported in peer-reviewed literature and confirmed by proposed qualitative research
Facilitators of PrEP use | Baseline
  7-item checklist of facilitators as previously reported in peer-reviewed literature and confirmed by proposed qualitative research
Injectable PrEP treatment modality preference | Baseline
  5- item Likert scale to report likelihood of using monthly injectable PrEP versus daily oral dosing
Implantable PrEP treatment modality preference | Baseline
  5- item Likert scale to report likelihood of using long-acting implantable PrEP versus daily oral dosing
Long-acting oral PrEP treatment modality preference | Baseline
  5- item Likert scale to report likelihood of using long-acting oral PrEP versus daily oral dosing
Intersectional anticipated discrimination scale | Baseline
  5-point Likert scale to measure likelihood of anticipated experiences with discrimination (subscale from Scheim and Bauer,2019; Intersectional Discrimination Index: 0-4 score for each of 11 items which are then averaged for a score of 0-4; higher mean score associated with greater risk of high risk sexual outcome as well as preference for long-acting PrEP treatment modalities that required less interaction with healthcare system)
Intersectional day-to-day discrimination index | Baseline
  4-point frequency scale to measure occurrence of day-to-day experiences with discrimination (subscale from Scheim and Bauer ,2019; Intersectional Discrimination Index: 0-2 score for each of 9 items for a range of values between 0-18; higher score associated with greater risk of high risk sexual outcome as well as preference for long-acting PrEP treatment modalities that required less interaction with healthcare system)
Intersectional major discrimination index | Baseline
  3-frequency scale for major experiences due to discrimination (subscale from Scheim and Bauer, 2019) Intersectional Discrimination Index: 0-2 score for each of 13 items which are then summed for scores of 0-26 (lifetime experience); higher scores associated with greater risk of high risk sexual outcome as well as preference for long-acting PrEP treatment modalities that required less interaction with healthcare system)

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel Dornsife School of Public Health, Philadelphia, Pennsylvania, United States